CLINICAL TRIAL: NCT03195114
Title: Multicenter Prospective CoreValve Study Using Cardiac MRI for Assessment of Paravalvular Aortic Regurgitation and Its Impact on LV Reverse Remodeling and Cardiovascular Outcomes
Brief Title: Cardiac MRI for Post-TAVR Paravalvular Leak Assessment
Acronym: Class-CMR
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Thomas Gleason, Associate Professor of Surgery, University of Pittsburgh
Other Study IDs: PRO15050330
Record Dates: First submitted 2017-03-12; First posted 2017-06-22 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Paravalvular Leak
Keywords: post TAVR quantification; cardiac MRI; echocardiography; biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Samples for future
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multimodality Imaging and Biomarkers: Post-TAVR patients who received commercial Medtronic Evolut-R or Evolut PRO bioprosthesis implant and found to have at least mild PVL on 1-month post-TAVR echocardiogram will undergo multimodality imaging and biomarkers evaluation at 1-month and 7-months post-TAVR.
  Interventions: Diagnostic Test: Multimodality Imaging and Biomarkers

INTERVENTIONS:
Diagnostic Test: Multimodality Imaging and Biomarkers — Cardiac MRI, Cardiac MDCT, Echocardiography and Biomarkers Testing

SUMMARY:
The objectives of this study are to: a) evaluate and correlate the severity of paravalvular leak (PVL) assessed by both cardiac MRI and transthoracic echocardiography (TTE) after transcatheter aortic valve replacement (TAVR) with Medtronic Evolut-R or Evolut PRO bioprostheses; b) assess the inter and intraobserver variability of both imaging methods; and c) correlate the severity of PVL with post-TAVR changes in LV remodeling and clinical outcomes.

DETAILED DESCRIPTION:
Paravalvular leak (PVL) represents the most common complication post-transcatheter aortic valve replacement (TAVR). Presence of even mild PVL has been associated with unfavorable outcomes including late mortality, which is physiologically and hemodynamically hard to be reconciled.

Although transthoracic echocardiogram (TTE) is the first line test for the PVL quantification, it can be flawed due to poor acoustic windows, eccentricity of PVL, image degradation associated with the implanted prosthesis, irregular orifices, subjectivity and inconsistency of the assessment and grading. Furthermore, to date, most published studies do not use a uniform standardized way of quantifying the PVL. The Valve Academic Research Consortium (VARC) published the VARC II definitions and suggested the use of TAVR-specific criteria for the assessment of PVL. However, there has been no validation of this proposed criteria and how their selected cutoffs correlate to patient outcomes. All these issues contribute to uncertainty and imprecision of the current method, leading to difficulties and subjectivity in the assessment and quantification of PVL severity.

Cardiac MRI (CMR) is able to directly quantify aortic regurgitation with high accuracy and reproducibility by using the technique of phase-contrast velocity mapping when compared to TTE. CMR had lower intraobserver and interobserver variabilities for regurgitant volume assessment, suggesting that CMR may be superior for serial measurements. In addition, CMR quantification of aortic regurgitant fraction allows risk-stratification identifying patients at risk for development of heart failure and need for aortic valve surgery.

However, despite these advantages, the use of CMR for PVL assessment post-TAVR has been limited. A recent single center prospective pilot study (n=16) showed that CMR assessment of PVL was feasible using CoreValve prosthesis. In addition, CMR rather than TTE, correlated better with intra-procedural aortography. TTE underestimated the degree of PVL compared to CMR suggesting the opportunity of this modality to more reliably and accurately quantify PVL after TAVR. Another recent small and single-center CMR study (n=43) compared immediate post-TAVI CMR findings with those at 6-month follow-up. There were 32 patients (74%) treated with Medtronic CoreValve prosthesis and 11 (26%) treated with Edwards Sapien XT valve. The authors noted significant favorable LV remodeling at 6 months, but not in patients with > mild PVL. Furthermore, PVL quantified by CMR did not decrease over time. Given the small number of patients, the authors could not compare the temporal changes between the two prosthesis. In addition, the mechanisms associated with the changes in PVL severity were not able to be ascertained given the study design.

CMR provides exquisite tissue characterization using late-gadolinium enhancement imaging. Adverse myocardial response to pressure-overload causes maladaptive myocardial hypertrophy with increased LV mass and also myocardial fibrosis (MF), which has been associated with adverse outcomes despite aortic valve replacement. Newer CMR techniques such as T1 mapping and extracellular volume fraction quantification can now non-invasively quantify the extent of diffuse MF supported by histological validation. The interplay between PVL and MF and their impact of on the LV reverse remodeling is unknown. It is possible that PVL might exert its detrimental effects by slowing LV reverse remodeling, hampering the regression of LV hypertrophy and myocardial fibrosis post-TAVR.

Lastly, gated multi-detector computed tomography (MDCT) which has a critical role in the pre-procedural planning of patients undergoing TAVR evaluation, also has been found important in identifying predictors of PVL post-TAVR. However, the role of MDCT in the post-TAVR setting, for PVL evaluation, has not been yet established. Gated MDCT post-TAVR might be relevant to determine the interplay between the native aortic valve/annulus and the TAVR prosthesis aiding in the evaluation of possible mechanism(s) behind PVL changes over time.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered for study participation if they meet all of the following inclusion criteria:

* Patient ≥ 60 years of age has undergone commercial TAVR implant with Evolut R or Evolut PRO bioprosthesis within prior 25-45 days.
* Patient has ≥ mild PVL on TTE study performed at approximately the one (1) month post-TAVR (regular clinical follow-up visit taking place within prior 25-45 days post-TAVR)
* The patient and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Eligible patients from the three (3) participating institutions (University of Pittsburgh, Pittsburgh, PA; Methodist Hospital, Houston, TX and Quebec Heart & Lung Institute, Quebec, Canada) who have received TAVR with Evolut R or Evolut PRO will be screened for this study. All patients should be willing and able to provide a written informed consent for this study.

Exclusion Criteria:

* Patients with unstable condition and/or with implanted permanent cardiac device such as implantable cardiac defibrillators, cardiac resynchronization device, etc. MRI-conditional pacemaker devices would not represent an exclusion given the proven safety of these devices at 1.5 Tesla magnetic field strength.
* Patients treated with valve-in-valve implantation technique to address moderate-severe PVL and/or prosthetic aortic valve dysfunction.
* Patients with significant interval cognitive decline post-TAVR, unable to follow instructions required for both MDCT and CMR studies.
* Patients with metallic objects or implanted medical devices in the body (i.e. non-MRI conditional cardiac pacemaker or defibrillator, central nervous system aneurysm clips,implanted neural stimulators, cochlear implant, ocular foreign body [e.g., metal shavings], other implanted medical devices [e.g., drug infusion port], insulin pump, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants) which would exclude the participant from participating in the study. Verification of safety for MRI study should be checked for each one of the implanted medical devices at the website www.mrisafety.com.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 55 men and women aged 60 or above who received Medtronic Evolut-R or Evolut PRO and have at least mild paravalvular leak on transthoracic echocardiogram performed 25-45 days after TAVR procedure.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
PVL severity regression | up to 7-months post-TAVR
  To test that PVL severity, assessed by CMR using regurgitant fraction and regurgitant volume, changes and regresses over a 6-month period post-TAVR (comparing those measurements at 1-month and 7-months post-TAVR).

SECONDARY OUTCOMES:
Intra- and inter-observer variability of PVL severity assessment | 1-month and 7-months post-TAVR
  To test the hypothesis that PVL severity, assessed by CMR using regurgitant fraction and regurgitant volume, at both 1-month and 7-months post-TAVR has lower intra and inter-observer variability when compared to its assessment by TTE.

OTHER OUTCOMES:
PVL severity change at 7-months post-TAVR is associated with LV mass regression and myocardial fibrosis | up to 7-months post-TAVR
  To test that PVL severity change by CMR over 6-month period post-TAVR (comparing assessment at 1-month vs 7-months post-TAVR regurgitant fraction and regurgitant volume), is a determinant of LV reverse remodeling and negatively correlates with the regression of LV mass and myocardial fibrosis assessed by CMR.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist DeBakey Heart & Vascular Center, Houston, Texas
- Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No